CLINICAL TRIAL: NCT05199597
Title: The Response to Atropine Drops (RAD) Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeffrey J. Walline, OD PhD, Associate Dean for Research, Ohio State University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021H0326
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Myopia
Keywords: atropine
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Participants will have one drop of low concentration atropine placed in one eye four different times in random order
Masking Description: The participant will not know which of the four drops is being administered in random order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants will receive all four drops in randomized order
  Interventions: Drug: 0.01% atropine; Drug: 0.05% atropine

INTERVENTIONS:
Drug: 0.01% atropine — 0.01%, room temp, Lab A
  Other Names: 0.01% atropine at room temperature from Lab A
Drug: 0.05% atropine — 0.05%, room temp, Lab A
  Other Names: 0.05% atropine at room temperature from Lab A
Drug: 0.05% atropine — 0.05%, refrigerated, Lab A
  Other Names: 0.05% atropine refrigerated from Lab A
Drug: 0.05% atropine — 0.05%, room temperature, Lab B
  Other Names: 0.05% atropine at room temperature from Lab B

SUMMARY:
The purpose of this study is to examine the comfort of giving low concentration atropine eye drops.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will answer questions about themselves and complete a 12-question survey about the need for drama. An examiner will then measure the sensitivity of the cornea (clear window on the front of the eye) by touching the cornea with a thin thread that shortens until it is first detected by the participant. After that, an examiner will place a drop of atropine in the right eye, and the participant will rate the eye comfort for 25 seconds using a computerized slide scale. Five minutes after the first drop, the examiner will put a drop in the left eye and the participant will rate the comfort for 25 seconds. The examiner will then repeat that process one more time with each eye. The drops placed in the eyes will be 0.01% atropine at room temperature from Lab A, 0.05% atropine at room temperature from Lab A, 0.05% atropine refrigerated from Lab A, or 0.05% atropine at room temperature from Lab B. The drops will be placed in the eyes in random order, so the participant won't know which one is being administered. At the very end, the participant will rate how likely s/he would be to take a low concentration atropine eye drop every day in each eye if it may delay the onset of nearsightedness from 1 (definitely not) to 10 (definitely would).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Time to Return to Baseline Comfort | We will record comfort of each drop for a maximum of 25 seconds
  We will compare the amount of time that it takes a participant to report that the eye comfort is "0," meaning that it returned to baseline comfort, for the following drop comparisons:
  1. 0.01% at room temperature from Lab A and 0.05% at room temperature from Lab A (comparing concentrations)
  2. 0.05% at room temperature from Lab A and 0.05% refrigerated from Lab A (comparing temperatures)
  3. 0.05% at room temperature from Lab A and 0.05% at room temperature from Lab B (comparing labs)

SECONDARY OUTCOMES:
Proportion Who Return to Baseline Comfort Within 25 Seconds | We will record comfort of each drop for a maximum of 25 seconds
  We will compare the proportion of participants who report the eye comfort is "0," meaning that it returned to baseline comfort, for the following drop comparisons:
  1. 0.01% at room temperature from Lab A and 0.05% at room temperature from Lab A (comparing concentrations)
  2. 0.05% at room temperature from Lab A and 0.05% refrigerated from Lab A (comparing temperatures)
  3. 0.05% at room temperature from Lab A and 0.05% at room temperature from Lab B (comparing labs) Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)
Peak Comfort Score | We will record comfort of each drop for a maximum of 25 seconds
  We will compare the peak comfort score, meaning the most discomfort, for the following drop comparisons:
  1. 0.01% at room temperature from Lab A and 0.05% at room temperature from Lab A (comparing concentrations)
  2. 0.05% at room temperature from Lab A and 0.05% refrigerated from Lab A (comparing temperatures)
  3. 0.05% at room temperature from Lab A and 0.05% at room temperature from Lab B (comparing labs) Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)
Average Comfort Score | We will record comfort of each drop for a maximum of 25 seconds
  We will compare the average comfort score over 25 seconds for the following drop comparisons:
  1. 0.01% at room temperature from Lab A and 0.05% at room temperature from Lab A (comparing concentrations)
  2. 0.05% at room temperature from Lab A and 0.05% refrigerated from Lab A (comparing temperatures)
  3. 0.05% at room temperature from Lab A and 0.05% at room temperature from Lab B (comparing labs) Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)
Correlation Between Peak Comfort Score and Corneal Sensitivity | We will record comfort of the drop for a maximum of 25 seconds
  We will determine the correlation coefficient between the peak pain score when taking 0.05% atropine at room temperature from Lab A and corneal sensitivity Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)
Correlation Between Peak Comfort Score and Iris Color | We will record comfort of the drop for a maximum of 25 seconds
  We will determine the correlation coefficient between the peak pain score when taking 0.05% atropine at room temperature from Lab A and iris color Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)
Correlation Between Peak Comfort Score and the Perceived Victim Scale Score | We will record comfort of the drop for a maximum of 25 seconds
  We will determine the correlation coefficient between the peak pain score when taking 0.05% atropine at room temperature from Lab A and the Persistent Perceived Victim scale score of the Need for Drama Survey Comfort scale ranges from 0 (no discomfort) to 10 (extreme discomfort)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
I do not plan to share the data